CLINICAL TRIAL: NCT01900626
Title: Single Versus Double Epidural Catheter Technique for Postoperative Analgesia Following Scoliosis Surgery
Brief Title: Single vs Double Epidural Catheter Analgesia for Scoliosis Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was unable to meet patient enrollment goals. PI chose to terminate the study early.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0109
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-04

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- single epidural catheter (Active Comparator)
  Interventions: Drug: epidural catheter
- double epidural catheter (Active Comparator)
  Interventions: Drug: epidural catheter

INTERVENTIONS:
Drug: epidural catheter — epidural catheter with 0.3% ropivacaine

SUMMARY:
This is a study comparing pain control utlilizing one or two epidural catheters, along with a hydromorphone PCA, for analgesia following surgery for correction of scoliosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery via a posterior approach for AIS
2. Children ages 11-18
3. ASA physical status 1-2
4. Informed consent by legal guardian and assent by patient (for minors 11-17 years of age) or informed consent by subject (for patients 18 years of age)
5. Planned correction of at least 8 vertebral levels

Exclusion Criteria:

1. Patient refusal to participate
2. Patients on chronic narcotic medication
3. Allergy to standard of care drugs used in the study (Omnipaque, ropivacaine, hydromorphone, oxycodone, acetaminophen, gabapentin, ondansetron, nalbuphine or diphenhydramine, diazepam)
4. Coagulopathy
5. Pre-existing neurological deficit
6. Inability to use a Numerical Rating Scale (NRS: 0-10 patient self-reported score) for pain assessment

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- American Family Children's Hospital, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 participants were enrolled in the study. However,this study was being closed due to difficulty with enrollment and changes to standard of care. No data was analysed for outcome measures.
Period: Overall Study
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — study was closed due to low enrollment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Epidural Catheter | Double Epidural Catheter | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores With Activity
Description: The pain scores will be examined using the Numeric Rating Scale (NRS). NRS score ranges from 0-10. Higher score represents more pain/worse outcome
Time Frame: 72 hours
Population: This study is being closed due to difficulty with enrollment and changes to standard of care. No participant data was collected for outcome measures
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pain Scores at Rest
Description: as for outcome 1
Time Frame: 72 hours
Population: as for outcome 1
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Opioid Usage
Description: Hydromorphone usage measured in mcg/kg/day. No min/max. More hydromorphone usage represents worse outcome
Time Frame: 72 hours
Population: This study is being closed due to difficulty with enrollment and changes to standard of care.No data analyses was done
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Outcomes:The Pediatric Outcomes Data Collection Instrument (PODCI) Score
Description: Functional outcome will be measured by the Pediatric Outcomes Data Collection Instrument (PODCI). Scores range from 0-100, lower score represents higher degree of disability
Time Frame: 3 months
Population: This study is being closed due to difficulty with enrollment and changes to standard of care.No data analyses was done
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Functional Outcomes: Scoliosis Research Society-22r (SRS-22r) Patient Questionnaire
Description: Functional outcome will be measured by the Scoliosis Research Society-22r (SRS-22r). Scores range from 0-110, higher scores represent less disability/better outcome
Time Frame: 3 months
Population: This study is being closed due to difficulty with enrollment and changes to standard of care.No data analyses was done
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Functional Outcomes: The Owestry Disability Index(ODI)
Description: Functional outcome will be measured by the Owestry Disability Index (ODI).
  ODI represents following disability levels:
  0% -20%: Minimal disability, 21%-40%: Moderate Disability, 41%-60%: Severe Disability, 61%-80%: Crippling back pain, 81%-100%: These patients are either bed-bound or have an exaggeration of their symptoms.
Time Frame: 3 months
Population: This study is being closed due to difficulty with enrollment and changes to standard of care.No data analyses was done
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This study is being closed due to difficulty with enrollment and changes to standard of care. No adverse event data was collected
Description: This study is being closed due to difficulty with enrollment and changes to standard of care.No adverse event data was collected
Groups:
- Single Epidural Catheter; Double Epidural Catheter: This study is being closed due to difficulty with enrollment and changes to standard of care. No data on serious adverse events was collected
Arm/Group | Single Epidural Catheter | Double Epidural Catheter
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes